CLINICAL TRIAL: NCT06168474
Title: Evaluating the Impact of a SIMPlified LaYered Consent Process on Recruitment of Potential Participants to the Staphylococcus Aureus Network Adaptive Platform Trial: a Pragmatic Nested Randomized Clinical Trial
Brief Title: Evaluating Simplified Layered Consent for Clinical Trials
Acronym: SIMPLY-SNAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Sean Ong, Research Associate, Evaluative Clinical Sciences, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 496741
Record Dates: First submitted 2023-11-23; First posted 2023-12-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: informed consent; research ethics; clinical trials; Staphylococcus aureus bacteremia; equity, diversity and inclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Neither study subjects nor research staff administering consent will be masked to intervention allocation, as masking of the two different consent processes is not feasible. However, to minimize bias in measurement of outcomes, the assessor of the secondary outcomes of participant satisfaction and understanding will not be directly involved in the consent process and will be masked to the intervention allocation. Analysis of outcome results will also be performed masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simplified layered consent process (Experimental): For participants randomized to the SIMPLY-SNAP experimental group, a simplified layered consent process will be used to explain information for the SNAP trial. The research staff member obtaining consent will provide a standardized explanation, providing summarized information in simple English or French contained in a 4-page concise participant information sheet. Throughout the consent process, the research staff member will answer any questions that the participant has, to reflect routine consent discussion practice.
  Interventions: Other: Simplified layered consent form
- Full-length consent form (Active Comparator): For participants randomized to the control group, the existing consent process will be used including going through the currently approved full-length informed consent form. The research staff member will provide an explanation using the full-length informed consent form as per standard clinical trial procedures. Similarly, throughout the consent process, the research staff member will answer any participant questions as per normal procedures.
  Interventions: Other: Full-length consent form

INTERVENTIONS:
Other: Simplified layered consent form — The simplified consent form includes all essential elements of trial consent including an explanation of the trial procedures, data and sample collection, and follow-up information. The form also outlines important ethical considerations for patients, such as confidentiality, regulatory and safety requirements, the ability to drop out, and the necessary process and contact numbers for grievances or feedback. In addition to the text, the form includes links to additional written information and videos that can be accessed on top of the simplified informed consent form (i.e., the additional layers in the layered consent process). These materials are hosted on the main SNAP trial website (https://www.snaptrial.com.au/patients) and are available in English and French. Participants will be able to access these directly through embedded hyperlinks using provided electronic tablets.
  Arms: Simplified layered consent process
Other: Full-length consent form — The full-length informed consent form contains all information upfront. Links to additional information will not be provided on the form but are freely available on the Internet should the participant wish to access them.
  Arms: Full-length consent form

SUMMARY:
The goal of this clinical trial (the SIMPLY-SNAP trial) is to compare a simplified layered consent form to a full-length consent form for use during the informed consent process for a larger clinical trial of treatment of Staphylococcus aureus bloodstream infection (the SNAP trial).

The main questions it aims to answer are:

* Does use of a simplified layered consent form lead to an increased recruitment rate to the SNAP trial?
* Does use of a simplified layer consent form lead to increased participant understanding of the SNAP trial and increased participant satisfaction with the informed consent process?

Participants will be randomized to either the full-length informed consent form or the simplified layered consent form containing links to optional supplementary information or videos. Research staff will use the assigned form to explain the SNAP trial to participants. After consent, participants will be evaluated on their understanding of the SNAP trial and satisfaction with the consent process using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All inclusion criteria from the larger SNAP trial:

  1. S. aureus complex grown from ≥1 blood culture
  2. Admitted to a participating hospital at the time of eligibility assessment
* Specific additional inclusion criteria for SIMPLY-SNAP:

  1. Admitted to participating hospital of SIMPLY-SNAP
  2. Self-reported proficiency in English or French adequate to be able to participate in consent process carried out solely in English or French (as the supplementary consent materials required in the simplified consent process are currently only available in these two languages)

Exclusion Criteria:

* All exclusion criteria from larger SNAP trial:

  1. Time of anticipated platform entry is greater than 72 hours post collection of the index blood culture
  2. Polymicrobial bacteremia, defined as more than one organism in the index blood cultures, excluding those organisms judged to be contaminants by either the microbiology laboratory or treating clinician
  3. Patient currently being treated with a systemic antibacterial agent that cannot be ceased
  4. Known previous participation in SNAP
  5. Known positive blood culture for S. aureus between 72 hours and 180 days prior to the time of eligibility assessment
  6. Treating team deems enrolment in the study is not in the best interest of the patient
  7. Treating team believes that death is imminent and inevitable
  8. Patient is for end-of-life care and antibiotic treatment is considered inappropriate
  9. Patient <18 years of age and paediatric recruitment not approved at recruiting site
* Specific additional exclusion criteria for SIMPLY-SNAP: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients recruited to SNAP | 1 day
  The number of patients who consented and were randomized in the SNAP trial, divided by the total number of patient eligible for the SNAP trial and randomized in SIMPLY-SNAP.

SECONDARY OUTCOMES:
Participant understanding of the clinical trial | Within 3 days after the consent process
  Understanding of the clinical trial will be measured by a modified Consent Understanding Evaluation (CUE) tool. This is a questionnaire that comprises a list of open and closed-ended questions designed to evaluate a participant's understanding of the clinical trial they just enrolled in. It is adapted from previous similar trials evaluating adjunctive consent interventions but modified to the context of SNAP. The score ranges from 0 (worst understanding) to 15 (best understanding).
Participant satisfaction with the consent process | Within 3 days after the consent process
  Scored by 11-point Likert scale (0 to 10; 0 being not satisfied at all and 10 being extremely satisfied).
Research staff satisfaction with the consent process | 1 day
  Scored by 11-point Likert scale (0 to 10; 0 being not satisfied at all and 10 being extremely satisfied).
Time taken for entire consent process | 1 day
  In minutes

OTHER OUTCOMES:
Diversity of enrolled trial population | End of the entire SIMPLY-SNAP study
  As an exploratory outcome, we will also evaluate diversity of the enrolled trial population across five self-reported socio-demographic characteristics: gender, ethnicity, primary spoken language, socioeconomic status (measured by income level, or last-income level before retirement), and highest formal educational level attained.
  We will separately evaluate diversity of the patient group enrolled in SNAP via the simplified consent process versus the patient group enrolled via the full-length consent form. Diversity will be measured using the Simpson's Diversity Index (SDI). SDI will be calculated for each of five socio-demographic variables for the group recruited via simplified consent and the group recruited via conventional consent. A composite diversity score for each group combining the SDIs of all five variables will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Sean WX Ong, MBBS, Principal Investigator — University of Toronto
Locations (6):
- Canada (6):
  - University of Calgary, Foothills Medical Centre, Peter Lougheed Centre, Rockyview Hospital, South Health Campus, Calgary, Alberta
  - Hamilton General Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ong SWX, Lee TC, Fowler RA, Mahar R, Pinto RL, Rishu A, Petrella L, Whiteway L, Cheng M, McDonald E, Johnstone J, Mertz D, Kandel C, Somayaji R, Davis JS, Tong SYC, Daneman N. Evaluating the impact of a SIMPlified LaYered consent process on recruitment of potential participants to the Staphylococcus aureus Network Adaptive Platform trial: study protocol for a multicentre pragmatic nested randomised clinical trial (SIMPLY-SNAP trial). BMJ Open. 2024 Jan 18;14(1):e083239. doi: 10.1136/bmjopen-2023-083239. PMID 38238170